CLINICAL TRIAL: NCT01185925
Title: PDE5-Inhibition With Sildenafil Reverses Exercise Oscillatory Breathing in Chronic Heart Failure: a Long-Term Cardiopulmonary Exercise Testing Placebo-Controlled Study
Brief Title: Exercise Oscillatory Breathing and Sildenafil in Heart Failure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Milan (Other)
Responsible Party: Marco Guazzi, Cardiopulmonary Unit, University of Milano
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 444-14; 14a
Record Dates: First submitted 2010-08-19; First posted 2010-08-20 (Estimated); Last update posted 2011-08-05 (Estimated); Status verified 2008-05

CONDITIONS: Heart Failure
Keywords: PDE5-inhibition; exercise ventilation; heart failure; sildenafil; pulmonary hemodynamics
MeSH Terms: conditions — Heart Failure | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Placebo (Placebo Comparator): Control Group
  Interventions: Drug: Placebo
- sildenafil, pde5 inhibitor (Active Comparator): treatment group; sildenafil 50 mg three times a day for 1 year
  Interventions: Drug: Sildenafil

INTERVENTIONS:
Drug: Sildenafil — Sildenafil, 50 mg 3 times/day
  Arms: sildenafil, pde5 inhibitor
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Exercise oscillatory breathing (EOB) is a ventilatory abnormality that occurs in approximately 20% of heart failure (HF) patients and carries a very unfavourable prognosis.

Pathophysiology seems quite complex and putative mechanisms include increased pulmonary capillary pressure and pulmonary vasoconstriction, circulatory blood-flow fluctuations in the pulmonary arterial system and instability of ventilatory control.

Inhibition of the phosphodiesterase 5 (PDE5) isoenzyme favourably regulates pulmonary vascular tone and permeability through over signaling of the endothelial nitric oxide pathway. The investigators tested the hypothesis that sildenafil would reverse the EOB pattern in patients with HF and pulmonary hypertension.

ELIGIBILITY:
Inclusion Criteria:

* consent to participate in the study after detailed information about benefits and risks
* negative exercise stress test prior to study initiation
* forced expiratory volume in 1 sec/forced vital capacity ratio >70%;
* LVEF < 45%.

Exclusion Criteria:

* inability to complete a maximal exercise test
* resting systolic blood pressure > 140 or <110 mmHg
* therapy with nitrate preparations
* history of sildenafil intolerance
* significant lung or valvular diseases
* neuromuscular disorders or peripheral vascular disease

Ages: 30 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2008-04; Primary Completion 2009-12 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Drug Effect on Oscillatory Breathing during Exercise | 1 year follow-up